CLINICAL TRIAL: NCT07138248
Title: Transvaginal Three-Dimensional Ultrasound in the Evaluation of Intrauterine Device Placement Six Weeks After Insertion: A Cross-Sectional Study
Brief Title: Transvaginal Three-Dimensional Ultrasound for Evaluation of Intrauterine Device Position Six Weeks After Insertion
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira khaled mohamed khafaga, Resident, Obstetric and Gynecology Department, Assiut University
Other Study IDs: TV3D-IUD-2025
Record Dates: First submitted 2025-08-16; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Evaluation of IUD Position Six Weeks After Insertion; Intrauterine Device Placement and Displacement
Keywords: Intrauterine Device; 3D Transvaginal Ultrasound; Postpartum Contraception

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postpartum Women Receiving IUD: Women aged 18-45 who undergo postpartum copper T380A IUD insertion, either vaginally or during cesarean delivery, and who consent to follow-up ultrasound at 6 weeks to assess IUD position.
  Interventions: Biological: 2D Transvaginal Ultrasound

INTERVENTIONS:
Biological: 2D Transvaginal Ultrasound — Three-dimensional transvaginal ultrasound used to assess the same outcomes as 2D, providing volumetric imaging and coronal reconstruction to detect displacement or malposition of the IUD

SUMMARY:
This study aims to evaluate the position of intrauterine devices (IUDs) six weeks after insertion using transvaginal three-dimensional (3D) ultrasound. Women aged 18-45 who undergo postpartum IUD insertion, either vaginally or during cesarean delivery, will be included. The study will compare the accuracy of 3D ultrasound versus conventional two-dimensional (2D) ultrasound in detecting IUD displacement, including partial expulsion, embedment, or perforation.

Participants will receive a copper T380A IUD, and all procedures will follow standard clinical protocols. Ultrasound assessments will be conducted six weeks after insertion to confirm proper placement. Data collected will include demographic information, reproductive history, and ultrasound findings.

The primary outcome is the prevalence of IUD displacement at six weeks. Secondary outcomes include the diagnostic accuracy of 3D versus 2D ultrasound. This study is designed to improve early detection of malpositioned IUDs, enhancing patient safety and contraceptive effectiveness.

DETAILED DESCRIPTION:
Intrauterine devices (IUDs) are highly effective, long-acting reversible contraceptives. Complications such as expulsion, perforation, and embedment can reduce contraceptive effectiveness and cause abnormal uterine bleeding or pelvic pain. Traditional 2D transvaginal ultrasound may fail to detect malpositioned IUDs, especially levonorgestrel-IUDs or when uterine anomalies are present. 3D transvaginal ultrasound offers improved visualization of the uterine cavity and IUD position.

Objectives

To evaluate the accuracy of 3D transvaginal ultrasound in detecting IUD displacement six weeks after insertion and compare it to conventional 2D ultrasound.

Methods

Study Design: Cross-sectional study Setting: Assiut General Hospital and Women's Health Hospital, Assiut, Egypt Duration: July 2025 - June 2026 Participants: Women aged 18-45 receiving postpartum IUD insertion (vaginal or cesarean) Sample Size: 138 women, accounting for 10% loss to follow-up

Procedures:

Participants provide written informed consent.

Baseline data collection: age, parity, residency, educational level, reproductive history, prior IUD use, dysmenorrhea, cervical surgery, lactation status.

Copper T380A IUD insertion:

Vaginal insertion: sterile technique, uterine sounding, insertion per manufacturer instructions.

Cesarean insertion: IUD placed in uterine fundus post-placenta delivery before uterine closure.

Follow-up at 6 weeks with 2D and 3D transvaginal ultrasound to assess IUD position.

Outcomes:

Primary: Prevalence of IUD displacement at 6 weeks

Secondary: Accuracy of 3D vs 2D ultrasound in detecting displacement, partial expulsion, embedment, and perforation.

Data Management:

Data entered and analyzed using SPSS v21.

Categorical variables: Chi-square or Fisher's exact test

Quantitative variables: Shapiro-Wilkes test for normality; Mann-Whitney or Student's t-test as appropriate

Significance: p < 0.05

Ethical Considerations

Study approved by Assiut Faculty of Medicine Ethical Review Committee

Conducted according to Declaration of Helsinki and Good Clinical Practice

Participant privacy and confidentiality ensured

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-45 years

Postpartum women receiving copper T380A IUD insertion, either vaginal or cesarean

Agree to participate and provide written informed consent

Exclusion Criteria:

* Uterine anomalies (e.g., bicornuate uterus)

Significant uterine pathology (e.g., large fibroids)

Puerperal sepsis

Refusal to insert IUD

Past history of IUD complications

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Postpartum women aged 18-45 undergoing copper T380A IUD insertion at Assiut General Hospital or Women's Health Hospital, Assiut, Egypt, who consent to follow-up ultrasound assessment six weeks after insertion.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of IUD displacement 6 weeks after insertion | 6 weeks after IUD insertion
  The proportion of postpartum women whose copper T380A IUD is malpositioned, partially expelled, embedded, or perforated as determined by transvaginal ultrasound at 6 weeks post-insertion

SECONDARY OUTCOMES:
Accuracy of 3D vs 2D transvaginal ultrasound in detecting IUD displacement | 6 weeks after IUD insertion
  Comparison of the diagnostic performance (sensitivity, specificity) of 3D versus 2D ultrasound in identifying malpositioned IUDs, including partial expulsion, embedment, or perforation
Accuracy of 3D vs 2D transvaginal ultrasound in detecting IUD displacement | 6 weeks after IUD insertion
  Comparison of the diagnostic performance (sensitivity, specificity) of 3D versus 2D ultrasound in identifying malpositioned IUDs, including partial expulsion, embedment, or perforation.

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Health Hospital, Assiut, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abuhamad AZ, Singleton S, Zhao Y, Bocca S. The Z technique: an easy approach to the display of the mid-coronal plane of the uterus in volume sonography. J Ultrasound Med. 2006 May;25(5):607-12. doi: 10.7863/jum.2006.25.5.607. PMID 16632784
- [Background] Benacerraf BR, Shipp TD, Bromley B. Three-dimensional ultrasound detection of abnormally located intrauterine contraceptive devices which are a source of pelvic pain and abnormal bleeding. Ultrasound Obstet Gynecol. 2009 Jul;34(1):110-5. doi: 10.1002/uog.6421. PMID 19565532
- [Background] Nosseir MA, et al. Role of 3D-Ultrasound in Patients with Abnormal Uterine Bleeding for Detection of IUCD Malposition. Benha Med J. 2024;41(4):1-9.
- [Background] Thonneau P, Goulard H, Goyaux N. Risk factors for intrauterine device failure: a review. Contraception. 2001 Jul;64(1):33-7. doi: 10.1016/s0010-7824(01)00215-3. PMID 11535211
- [Background] Benacerraf BR, Shipp TD, Lyons JG, Bromley B. Width of the normal uterine cavity in premenopausal women and effect of parity. Obstet Gynecol. 2010 Aug;116(2 Pt 1):305-310. doi: 10.1097/AOG.0b013e3181e6cc10. PMID 20664389
- [Background] Wildemeersch D, Pett A, Jandi S, Hasskamp T, Rowe P, Vrijens M. Precision intrauterine contraception may significantly increase continuation of use: a review of long-term clinical experience with frameless copper-releasing intrauterine contraception devices. Int J Womens Health. 2013 Apr 30;5:215-25. doi: 10.2147/IJWH.S42784. Print 2013. PMID 23658502
- [Background] Teal SB, Sheeder J. IUD use in adolescent mothers: retention, failure and reasons for discontinuation. Contraception. 2012 Mar;85(3):270-4. doi: 10.1016/j.contraception.2011.07.001. PMID 22067773
- [Background] Lopez LM, Bernholc A, Zeng Y, Allen RH, Bartz D, O'Brien PA, Hubacher D. Interventions for pain with intrauterine device insertion. Cochrane Database Syst Rev. 2015 Jul 29;2015(7):CD007373. doi: 10.1002/14651858.CD007373.pub3. PMID 26222246
- [Background] Goldstuck ND, Wildemeersch D. Role of uterine forces in intrauterine device embedment, perforation, and expulsion. Int J Womens Health. 2014 Aug 7;6:735-44. doi: 10.2147/IJWH.S63167. eCollection 2014. PMID 25143756
- [Background] Committee on Practice Bulletins-Gynecology, Long-Acting Reversible Contraception Work Group. Practice Bulletin No. 186: Long-Acting Reversible Contraception: Implants and Intrauterine Devices. Obstet Gynecol. 2017 Nov;130(5):e251-e269. doi: 10.1097/AOG.0000000000002400. PMID 29064972